CLINICAL TRIAL: NCT04447547
Title: Clinical Trial of SL1904B CAR-T Cells for Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Collaborators: Beijing Lu Daopei Hospital (Other); Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1904B for NHL
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-08

CONDITIONS: Non-hodgkin's Lymphoma
Keywords: NHL，CD19
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SL1904B CAR-T (Experimental): Patients will be treated with CD19 CAR-T cells
  Interventions: Biological: CD19 CAR-T

INTERVENTIONS:
Biological: CD19 CAR-T — Biological: CD19 CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis;

SUMMARY:
This is a study of patients with relapsed or refractory non-Hodgkin's lymphoma. To evaluate the safety and efficacy of SL1904B in patients with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
The CARs consist of an anti-CD19 single-chain variable fragment（scFv） that was derived from the FMC63 mouse hybridoma, a portion of the human CD137（4-1BB） molecule, and the intracellular component of the human CD3ζ molecule. Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

The Main research objectives:

To evaluate the safety and efficacy of SL1904B in patients with recurrent or refractory non-Hodgkin's lymphoma

The Secondary research objectives:

To investigate the cytokinetic characteristics of SL1904B in patients with recurrent or refractory non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form and be willing and able to comply with the visit, treatment regimen, laboratory examination and other requirements of the study as stipulated in the trial flow chart;
2. The diagnosis of patients with relapsed or refractory non-hodgkin lymphoma;
3. There should be at least one measurable tumor focus according to the RECIST version 1.1;
4. ECOG Scores: 0~2;
5. The expression of CD19 on the tumor cells was reported as positive by either immunohistochemistry or flow cytometry;
6. Estimated survival time was longer than 3 months;
7. main organ functions shall meet the following requirements including: serum creatinine ≤1.5 times the upper limit of normal value (ULN); ALT ULN 2.5 or less; AST ULN 2.5 or less; Total bilirubin ≤ 1.5ULN; Left ventricular ejection fraction (LVEF) ≥45%; Hemoglobin ≥90g/L; Platelet count ≥50×109/L; absolute Neutrophil count (ANC) ≥1.0×109/L; Blood oxygen saturation >92%；
8. Peripheral blood mononuclear immune cells must be collected at least 2 weeks after the last radiotherapy or systemic treatment.

Exclusion Criteria:

1. Serious cardiac insufficiency；
2. Has a history of severe pulmonary function damaging;
3. With other tumors which is/are in advanced malignant and has/have systemic metastasis;
4. Merging the metabolic diseases (except diabetes);
5. Merging severe autoimmune diseases or immunodeficiency disease;
6. Patients with active hepatitis B or hepatitis C virus infection;
7. Patients with HIV infection or syphilis infection;
8. Has a history of serious allergies on Biological products (including antibiotics);
9. Participated in any other clinical drug trial for the last six months;
10. Being pregnant and lactating or having pregnancy within 12 months;
11. With other uncontrolled diseases and considered not suitable to participate by the researchers;
12. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within first one month after SL1904B infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Overall Remission Rate (ORR) | 3 months post CAR-T cells infusion
  Overall Remission Rate (ORR) including partial remission and complete remission rate after infusion of SL1904B

SECONDARY OUTCOMES:
Efficacy:duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD19 CAR- T cells in the genomes of PBMC by qPCR method and percentage of CD19 CAR- T cells measured by flow cytometry method
Cytokine release | First month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD&MD, Principal Investigator — Beijing Lu Daopei Hospital
Locations (2):
- China (2):
  - BeiJing Ludaopei Hospital, Beijing, Yizhuang
  - He bei Yan da Lu dao pei Hospital, Yanda